CLINICAL TRIAL: NCT02929576
Title: A Phase 3, Randomized, International Study Comparing the Efficacy and Safety of Enzalutamide in Combination With Paclitaxel Chemotherapy or as Monotherapy Versus Placebo With Paclitaxel in Patients With Advanced, Diagnostic-Positive, Triple-Negative Breast Cancer
Brief Title: Efficacy and Safety Study of Enzalutamide in Combination With Paclitaxel Chemotherapy or as Monotherapy Versus Placebo With Paclitaxel in Patients With Advanced, Diagnostic-Positive, Triple-Negative Breast Cancer
Acronym: ENDEAR
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Further understanding about the role of androgen signaling in TNBC was required
Sponsor: Pfizer (Industry)
Collaborators: Astellas Pharma Inc (Industry); Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MDV3100-20; 2016-000796-25 (EudraCT Number)
Record Dates: First submitted 2016-09-07; First posted 2016-10-11 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Breast Cancer
Keywords: metastatic; triple negative
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — enzalutamide; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Double-blind enzalutamide with paclitaxel (Experimental)
  Interventions: Drug: Enzalutamide; Drug: Paclitaxel
- Double-blind placebo with paclitaxel (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Paclitaxel
- Open-label enzalutamide monotherapy followed by paclitaxel (Experimental): At the time of disease progression, enzalutamide treatment will be discontinued and paclitaxel will be administered if considered to be an appropriate treatment by the treating physician until second disease progression.
  Interventions: Drug: Enzalutamide; Drug: Paclitaxel

INTERVENTIONS:
Drug: Enzalutamide — Enzalutamide will be administered as four 40-mg capsules once daily (160 mg/day).
  Other Names: Xtandi; MDV3100
  Arms: Double-blind enzalutamide with paclitaxel; Open-label enzalutamide monotherapy followed by paclitaxel
Drug: Placebo
  Arms: Double-blind placebo with paclitaxel
Drug: Paclitaxel — Paclitaxel (90 mg/m2) will be administered by constant-rate intravenous infusion of ≤ 1 hour once weekly for 16 weeks. Dose reductions or alterations to the schedule are allowed to maintain patient safety.

SUMMARY:
The purpose of this study is to evaluate and compare the clinical benefit and safety of treatment with enzalutamide in combination with paclitaxel chemotherapy or as monotherapy versus placebo with paclitaxel in patients with locally advanced or metastatic, diagnostic-positive, triple-negative breast cancer (TNBC).

ELIGIBILITY:
Inclusion Criteria:

* Adult women and men at least 18 years of age and willing and able to provide informed consent.
* Has advanced TNBC:
* TNBC is defined as staining by immunohistochemistry (IHC) < 1% or Allred score < 2 for estrogen receptor (ER) and progesterone receptor (PgR), and 0 or 1+ by IHC for human epidermal growth factor receptor 2 (HER2) or negative for gene amplification (average HER2 copy number < 4 signals/cell; HER2:CEP17 ratio < 2.0).
* Advanced disease is defined as locally advanced or metastatic disease not amenable to curative intent surgery or radiotherapy.
* Has diagnostic-positive status as determined by a central diagnostic testing laboratory.
* Received 0 or 1 prior line of systemic therapy in the advanced disease setting.
* Patients who received 1 prior line of therapy for locally advanced or metastatic TNBC must have objective disease progression as assessed by the investigator.
* Has measurable and/or disease that is not measurable but is evaluable using RECIST 1.1 (eg, bone metastases, pathologic lymph nodes, or skin lesions).
* Patients with nonmeasurable and nonevaluable TNBC (eg, malignant effusions or bone marrow as the only manifestations of disease) are not eligible for enrollment.
* Patients with metastatic disease limited to the bone must have disease adequately visualized by computed tomography (CT) with bone windows, magnetic resonance imaging (MRI), or x-ray.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1 at screening and a life expectancy of at least 3 months from randomization.

Exclusion Criteria:

* Received a taxane regimen ≥ 28 days in duration in the advanced disease setting.
* Prior taxane therapy for neoadjuvant and/or adjuvant disease is permitted.
* A single dose of a taxane given as part of an every-3-weeks regimen is permitted.
* Two doses of a taxane given as part of a once-weekly regimen is permitted.
* Had a disease-free interval of ≤ 12 months from the last dose of taxane when used as part of adjuvant therapy for patients who did not receive prior therapy for locally advanced or metastatic breast cancer.
* Has history of or known central nervous system (CNS) metastasis or active leptomeningeal disease; brain imaging is required for all patients during screening.
* Received any anticancer agent (commercially available or investigational) within 14 days before randomization.
* Received treatment with any of the following medications within 14 days before randomization:
* Estrogens, including hormone replacement therapy
* Androgens (eg, testosterone, dehydroepiandrosterone)
* Systemic radionuclides (eg, samarium, strontium)
* Had major surgery within 4 weeks before randomization.
* Has a history of another invasive cancer within 3 years before randomization, with the exception of fully treated cancers with a remote probability of recurrence.
* Has a history of a seizure condition or any condition that may predispose to seizure (eg, prior cortical stroke or significant brain trauma).
* Has known hypersensitivity to any of the enzalutamide/placebo capsule components.
* Had a hypersensitivity reaction to Cremophor EL (polyoxyethylated castor oil) or a drug formulated in Cremophor EL, such as paclitaxel, unless successfully treated and rechallenged with appropriate premedications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Anticipated in about 31 months following first patient enrolled

SECONDARY OUTCOMES:
Overall survival | Anticipated in about 40 months following first patient enrolled
PFS assessed by the investigator using Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 | Anticipated in about 31 months following first patient enrolled
Time to treatment failure | Anticipated in about 31 months following first patient enrolled
Best overall response | Anticipated in about 31 months following first patient enrolled
  Best overall response is defined as the best tumor response (complete response [CR], partial response [PR], stable disease, progressive disease, not evaluable) based on investigator assessment per RECIST 1.1 over all tumor assessments performed any time on study. Best objective response rate is defined as the proportion of patients with a best overall response of CR or PR for all patients based on investigator assessment per RECIST 1.1. The 2-sided 95% Confidence Interval (CI) will be reported for each treatment group using the Clopper-Pearson method.
Duration of response | Anticipated in about 31 months following first patient enrolled
Time to second disease progression in patients randomly assigned to enzalutamide monotherapy who subsequently receive paclitaxel | Anticipated in about 31 months following first patient enrolled
Clinical benefit rate at 24 weeks (CBR24): From the start of treatment D1 assessed every 8 weeks +/- 1 week while on study treatment | 24 weeks
  CBR (complete, partial response, or stable disease lasting 24 weeks or longer) assessed per RECIST 1.1
Safety as assessed by percentage of patients with any Adverse Event (AE), AE leading to Study Drug Discontinuation, AE leading to death, Serious Adverse Event (SAE), AE related to study drug, SAE related to study drug | Anticipated in about 31 months following first patient enrolled
Time to functional status deterioration using the Functional Assessment of Cancer Therapy-Breast (FACT-B) trial outcome index (physical, functional, breast) (TOI-PFB) | Anticipated in about 31 months following first patient enrolled
Pharmacokinetics of enzalutamide as assessed by trough plasma concentrations | Anticipated in about 31 months following first patient enrolled
Pharmacokinetics of the active metabolite N-desmethyl enzalutamide as assessed by trough plasma concentrations | Anticipated in about 31 months following first patient enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (6):
  - Topeka, Kansas
  - Metairie, Louisiana
  - The Bronx, New York
  - Houston, Texas
  - Tacoma, Washington
  - Wenatchee, Washington

IPD SHARING:
Plan to Share IPD: No